CLINICAL TRIAL: NCT04858945
Title: Using Teach Back to Improve Postpartum Maternal-infant Health Among Women With Limited Maternal Health Literacy: A Randomized, Controlled Study
Brief Title: Using Teach Back to Improve Postpartum Maternal-infant Health Among Women With Limited Maternal Health Literacy
Acronym: TB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Aalto University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CGZ-01
Record Dates: First submitted 2021-04-14; First posted 2021-04-26 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Pregnant Women
Keywords: maternal; health literacy; Postpartum Period; Health; Infant; Educational Technology

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach-back group (Experimental): The first education session will be arranged at the day or the following day of admission before delivery, with a group meeting involving three women and one educator. The main purpose of the first session is to help women understand and prepare for the labor. On the day of discharge after delivery, women will receive the second group education session hosted by an educator. The main purpose of the second session is to help women understand postpartum health issues, get to know the practice of postpartum recovery and learn newborn care skills. At two-week postpartum, a short online meeting will be arranged. During the meeting, the educator answers questions raised by the woman and gives advices on the challenges and difficulties in postpartum recover and caring newborn faced by the woman.
  Interventions: Behavioral: Teach-back method
- Control group (Active Comparator): Teach-back group and control group share some education content and communication methods, e.g. power-point presentation, educational video clips, live demonstration, information booklet, group discussion, and Q&A, expect that before the end of each education session.
  Interventions: Behavioral: Teach-back method

INTERVENTIONS:
Behavioral: Teach-back method — During the trial, women from teach-back group and controlled group will receive three education sessions The topics discussed at the first session included delivery mode, labor process and pain relief, newborn health and care (common health issues and care skills), perinatal die and excises, and perinatal psychological health. The topics discussed at the second session includ postpartum recovery, postpartum maternal health, perineum care (diet, oral care, perineal care, and hygiene), breastfeeding, postpartum blue and depression, neonatal care, neonatal screening tests, newborn vaccination and early child development. At two-week postpartum, the educator answers questions raised by the woman and gives advices on the challenges and difficulties in postpartum recover and caring newborn faced by the woman.

SUMMARY:
This is a randomized controlled trial study with two arms teach-back group vs. controlled group. We decided the assignment of the women to each group by tossing a coin (heads for the teach-back group and tails for the control group). The women were informed about receiving education during the trial, but they were not aware of the forms and techniques used in the trial, nor were they aware if they were assigned to the teach-back group or control group. For the first two education sessions, the women were grouped based on the time of their recruitment, i.e., being the first recruited, being the first grouped and being the first to receive education. The educators were numbered from 1 to 8 according to their work shifts and were assigned to education sessions in sequence and cycle. For the third education session, the educators were assigned to contact women based on the matching of their work schedules. The women could be grouped with different peers and met different educators during the trial. In this way, we could reduce the possible influence of educators and group peers on the results of the trial.

DETAILED DESCRIPTION:
Education for teach-back group and control group During the trial, women from teach-back group and controlled group will receive three education sessions arranged by trained nursing supervisors who played the educator role. The first education session is arranged at the day or the following day of admission before delivery, with a group meeting involving three women and one educator. The main purpose of the first session is to help women understand and prepare for the labor. The topics discussed at the first session includ delivery mode, labor process and pain relief, newborn health and care (common health issues and care skills), perinatal die and excises, and perinatal psychological health. On the day of discharge after delivery, women will receive the second group education session hosted by an educator. The main purpose of the second session is to help women understand postpartum health issues, get to know the practice of postpartum recovery and learn newborn care skills. The topics discussed at the second session includ postpartum recovery, postpartum maternal health, perineum care (diet, oral care, perineal care, and hygiene), breastfeeding, postpartum blue and depression, neonatal care, neonatal screening tests, newborn vaccination and early child development. At two-week postpartum, a short online meeting will be arranged between one woman and one educator. During the meeting, the educator answer questions raised by the woman and give advices on the challenges and difficulties in postpartum recover and caring newborn faced by the woman. teach-back group and control group share same education content and communication methods, e.g. power-point presentation, educational video clips, live demonstration, information booklet, group discussion, and Q&A, expect that before the end of each education session, women in teach-back group will be asked to use their own words to restate what was just learned and the educator assesses the patient's understanding of the subject, identifies misunderstandings, corrects the mistaken, and provides additional information if required until women can correctly restate what they were expected to learn.

ELIGIBILITY:
Inclusion Criteria:

1. over 18 years of age;
2. basically healthy and without being diagnosed with pregnancy complications;
3. with sufficient commands of communication in Chinese ;
4. at the pregnancy week between 37+0 and 41+6 but having no sign of labor or getting into the first stage of labor;
5. obtaining 27 or less points in the baseline measurement of MHL using perinatal maternal health literacy scale.

and Newborns who were :

1. born between 37 and 42 weeks of gestation age;
2. having a minimum apgar score of 8 after 5 minutes of being born;
3. with birth weights between 2500g and 4000g.

Exclusion Criteria:

1. women suffered from severe perinatal complications which required advanced special care e.g. transferring to intensive care unit (ICU)
2. fetal congenital malformations were diagnosed during the trial
3. women did not completed any of the required education sessions planned in the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
Maternal Health Literacy | Change from Baseline PMHLS at postpartum 42 days
  Perinatal Maternal Health Literacy Scale (PMHLS) To measure women's MHL at baseline (on the day when women just admitted to hospital) and 42 days postpartum, we employ perinatal maternal health literacy scale (PMHLS) that was brought up and validated in 2014 by a research team from Central South University in China [54]. PMHLS was developed by reference to the 55 knowledge and skill items defined in "Maternal and child health literacy - basic knowledge and skills", a national guidebook issued by China Ministry of Health in 2012 [55], which was also used by this study as the key source of developing educational interventions for both groups. PMHLS is comprised of 34 items with two response categories (correct =1, error/unknown=0). The range of total score is from 0 to 34, higher score indicating a higher level of maternal health literacy. The cut off score is 27, which means that women obtaining 27 points or less are deemed to be with low or limited maternal health literacy.
Postpartum health behaviours | up to postpartum 42 days
  Exclusive breastfeeding 24 hours postpartum,exclusive breastfeeding 42 days postpartum,uptake at the 42 days postpartum check-up,complete uptake of recommended vaccines
Maternal-infant health outcomes | up to postpartum 42 days
  Postpartum infection,subinvolution of uterus,acute mastitis,postpartum constipation,overweight,diaper dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Guizhi Cheng, Study Chair — Anhui Provincial Hospital
Locations (1):
- the First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
The dataset generated and analysed for this study is not publicly available due to the restrictions claimed in the document of the research permission and ethical approval. But the data are available from the ethics committee of the First Affiliated Hospital Ethics Committee of USTC for researchers who meet the criteria for access to confidential data. To request access to the data, please contact the ethics committee of the First Affiliated Hospital Ethics Committee of USTC or the main researcher Qianqian Ni.

REFERENCES:
- [Derived] Cheng GZ, Chen A, Xin Y, Ni QQ. Using the teach-back method to improve postpartum maternal-infant health among women with limited maternal health literacy: a randomized controlled study. BMC Pregnancy Childbirth. 2023 Jan 9;23(1):13. doi: 10.1186/s12884-022-05302-w. PMID 36624440